CLINICAL TRIAL: NCT01473745
Title: The Nasal Changes Affected by 2 Different Alar Base Suture Techniques After Maxillary LeFort I Osteotomy--A Randomized Controlled Trial
Brief Title: The Nasal Changes Affected by Different Alar Base Suture Techniques After Maxillary LeFort I Osteotomy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CGMH-100-1653A3; ChangGungMH (Other: ChangGungMH)
Record Dates: First submitted 2011-11-15; First posted 2011-11-17 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2011-08

CONDITIONS: Conditions in T74.31 or T76.31
Keywords: Alar Base Suture; Nasolabial Change; 3D stereogrammetry

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- modified alar base cinch suture (Active Comparator): Before closure of the maxillary wound, an alar base cinch suture was performed with 3-O Nylon. The modified alar cinch suture began from the bilateral alar part of the nasalis muscle and dermis tissue over the alar base, and then passed through a hole drilled on the anterior nasal spine.
  Interventions: Procedure: modified alar base cinch
- conventional alar base cinch suture (Placebo Comparator): Before closure of the maxillary wound, an alar base cinch suture was performed with 3-O Nylon. The conventional alar base cinch suture began from the bilateral alar part of the nasalis muscle and passed through a hole drilled on the anterior nasal spine.
  Interventions: Procedure: conventional alar base cinch

INTERVENTIONS:
Procedure: conventional alar base cinch — The conventional suture began from the bilateral alar part of the nasalis muscle and passed through a hole drilled on the anterior nasal spine.
  Other Names: conventional alar cinch suture technique
  Arms: conventional alar base cinch suture
Procedure: modified alar base cinch — The modified suture began from the bilateral alar part of the nasalis muscle and dermis tissue over the alar base, and then passed through a hole drilled on the anterior nasal spine.
  Other Names: modified alar base cinch technique
  Arms: modified alar base cinch suture

SUMMARY:
study hypothesis

1. The aim of this study:

   How can the investigators predict and control the nasal changes after maxillary LeFort I osteotomy with 2 different alar base suture techniques ?
2. Study hypothesis

   * Null hypothesis: Nasal changes were not affected by 2 different alar base suture techniques after maxillary LeFort I osteotomy
   * Alternative : Nasal changes were affected by 2 different alar base suture techniques after maxillary LeFort I osteotomy

DETAILED DESCRIPTION:
Background and study purpose:

Patients who received maxillary LeFort I osteotomy often complained about their nose become wider and more nostril show after surgery. According the the literature review, the conventional and modified alar base cinch technique both could control the interalar width. However, there is no long term result show which technique is superior to the other. Therefore, in order to improve patients' nasal and midfacial esthetics after the surgery, this study is to evaluate how the nasal changes affected by 2 different alar base cinch suture and which technique could result in a more positive effect.

ELIGIBILITY:
Inclusion Criteria:

* Taiwanese patients who received LeFort I osteotomy at CGMH during 2011-2012
* No previous craniofacial surgery
* Patients agreed to attend this study and willing to sign the agreement
* Patients who are elder than 18 years old and after growth completion

Exclusion Criteria:

* Craniofacial anomalies
* cleft lip and /or palate patients
* patients without all the documents
* patients do not receive combined correcting nasolabial shape and orthognathic surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-07; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen, Wen Ching Ko, DDS,MS, Study Director — Chang Gung MH; YiHsuan Chen, DDS, MS, Principal Investigator — Chang Gung MH
Locations (1):
- Chang Gung memorial hospital, Taipei, Taiwan, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All nongrowing Taiwanese patients over 18 years of age who underwent LeFort I maxillary osteotomy to correct skeletal discrepancies were randomly selected to receive either conventional or modified alar base cinching during the intraoral wound closing procedure.The recruitment duration was September of 2011 to February of 2013.
Pre-assignment Details: Exclusion criteria: Patients with an associated syndromic diagnosis, cleft of the lip or palate, dentofacial trauma, and previous nasal septum or nasal tip operations. 10 non-Class III patients were further excluded for enhanced sample consistency, 2 patients refused to participate were also excluded. Thus, total sample size was 48 patients.
Groups:
- Conventional Alar Cinch Group: Patients received conventional alar base cinch technique during LeFort I osteotomy procedure.
- Modified Alar Cinch Group: Patients received modified alar base cinch technique during LeFort I osteotomy procedure.
Period: Overall Study
Arm/Group | Conventional Alar Cinch Group | Modified Alar Cinch Group
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Taiwanese Class III patients
Groups:
- Modified Alar Cinch Suture: modified extraoral alar cinch suture techniques suture from intraoral to extraoral and from one side to another side
  modified extraoral alar base cinch technique: modified alar cinch suture technique performed after the maxillary Lefort I osteotomy.
- Conventional Alar Base Cinch Suture: conventional nasal cinch alar base technique: suture goes through bilateral alar base and anterior nasal spine(ANS) intra-orally
  conventional nasal alar cinch suture technique: conventional alar cinch suture technique performed after the maxillary Lefort I osteotomy.
- Total: Total of all reporting groups
Arm/Group | Modified Alar Cinch Suture | Conventional Alar Base Cinch Suture | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Customized [Mean (Full Range); unit: years]
  Age | 24.13 [19 to 57] | 23.78 [18 to 34] | 23.92 [18 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 7 | 6 | 13
Race/Ethnicity, Customized [Number; unit: participants]
  Taiwanese | 24 | 24 | 48
Region of Enrollment [Number; unit: participants]
  Taiwan | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Soft and Hard Tissue Landmarks Movement
Description: The investigator measured the movement (1 month minus baseline) of hard tissue landmarks before and after 4-6 weeks maxillary LeFort I osteotomy. The movement (6 months minus baseline) of soft tissue landmarks was measured before and after 6 months of the maxillary LeFort I osteotomy.
  The 3D directional movement of each point was measured in the x(transverse), y(vertical), and z (antero-posterior)planes. The positive directional movement of each point in X axis means the point moved left after surgery, and negative directional movement in X axis means the the point moved right after surgery. The positive directional movement in Y axis means the point moved upward after surgery, and negative directional movement in Y axis means the the point moved downward after surgery. The positive directional movement in Z axis means the point moved anteriorly after surgery, and negative directional movement in Z axis means the the point moved posteriorly after surgery.
Time Frame: The hard tissue movements were assessed after surgery 4-6 weeks.The soft tissue movements were assessed after surgery 6 months.
Population: similar sex distribution in both groups (7 male and 17 female patients in Group C, and 8 male and 16 female patients in Group M)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Modified Alar Cinch Suture | Conventional Alar Base Cinch Suture
Number analyzed (Participants) | 24 | 24
mm
  ANS point X axis | 0.95 (1.29) | -0.5 (1.09)
  ANS point Y axis | -0.95 (2.10) | -0.32 (2.82)
  ANS point Z axis | 0.50 (2.35) | -0.71 (2.73)
  A point X axis | 0.22 (1.50) | -0.58 (1.22)
  A point Y axis | -1.58 (1.95) | -0.95 (2.29)
  A point Z axis | 1.11 (2.43) | 1.83 (2.97)
  UI level X axis | -0.86 (1.53) | 0.30 (1.44)
  UI level Y axis | -1.08 (1.82) | -0.58 (2.40)
  UI level Z axis | 2.42 (3.95) | 1.91 (2.88)
  pronasale X axis | -0.35 (1.70) | 0.14 (1.23)
  pronasale Y axis | -0.29 (1.42) | -0.12 (1.62)
  pronasale Z axis | 0.48 (1.04) | 0.08 (1.43)
  subnasale X axis | -0.67 (1.88) | 0.05 (1.13)
  subnasale Y axis | -0.62 (1.32) | 0.21 (0.97)
  subnasale Z axis | 1.08 (1.89) | -0.03 (1.55)
  labiale suprious X axis | -0.74 (2.02) | 0.00 (1.64)
  labiale suprious Y axis | -0.03 (2.09) | -0.90 (1.78)
  labiale suprious Z axis | -0.03 (2.09) | 0.42 (2.06)
Statistical Analysis 1: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; ANS X axis; Test type: Superiority or Other; p = 0.098, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 2: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; ANS Y axis; Test type: Superiority or Other; p = 0.389, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 3: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; ANS Z axis; Test type: Superiority or Other; p = 0.780, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 4: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; A point X axis; Test type: Superiority or Other; p = 0.054, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 5: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; A point Y axis; Test type: Superiority or Other; p = 0.323, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 6: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; A point X axis; Test type: Superiority or Other; p = 0.371, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 7: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; UI level X axis; Test type: Superiority or Other; p = 0.011, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 8: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; UI level Y axis; Test type: Superiority or Other; p = 0.426, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 9: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; UI level Z axis; Test type: Superiority or Other; p = 0.621, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 10: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; pronasale X axis; Test type: Superiority or Other; p = 0.275, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 11: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; pronasale Y axis; Test type: Superiority or Other; p = 0.361, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 12: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; pronasale Z axis; Test type: Superiority or Other; p = 0.284, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 13: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; subnasale X axis; Test type: Superiority or Other; p = 0.119, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 14: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; subnasale Y axis; Test type: Superiority or Other; p = 0.019, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 15: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; subnasale Z axis; Test type: Superiority or Other; p = 0.034, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 16: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; labiale superious X axis; Test type: Superiority or Other; p = 0.422, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 17: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; labiale superious Y axis; Test type: Superiority or Other; p = 0.177, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 18: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; labiale superious Z axis; Test type: Superiority or Other; p = 0.133, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)

2. Secondary Outcome: 14 Nasolabial Linear Parameters
Description: 1. baseline characteristics: intercanthulus distance
  2. nasal linear parameters
  3. nasolabial linear parameters
Time Frame: up to post-operation 6 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Modified Alar Cinch Suture | Conventional Alar Base Cinch Suture
Number analyzed (Participants) | 24 | 24
mm
  Intercanthal distance change | 0.04 (0.82) | -0.62 (2.35)
  nasal height change | 0.78 (2.27) | -0.80 (3.91)
  nasal length change | 0.38 (2.41) | -0.81 (2.88)
  nasal tip protrusion change | -0.11 (0.92) | 0.46 (1.42)
  Nasal width change | 0.31 (1.31) | 0.13 (2.25)
  Alar base width change | 0.62 (2.08) | 0.26 (1.85)
  R nostril show vertical dimension change | -0.19 (1.52) | -0.27 (1.21)
  L nostril show vertical dimension | -0.20 (1.42) | -0.13 (1.87)
  Columellar length change | 0.38 (1.92) | 0.97 (1.60)
  Cutaneous height of upper lip change | 0.81 (1.87) | 0.38 (1.11)
  Overall upper lip height change | 0.63 (1.50) | 0.25 (1.86)
  Vermilion height of upper lip change | 0.55 (1.64) | 0.55 (1.35)
  Lower prolabial width change | -0.76 (1.56) | -0.40 (1.61)
  Upper lip protrusion change | -1.88 (3.26) | 0.41 (5.12)
Statistical Analysis 1: Comparison: Conventional Alar Base Cinch Suture; Intercanthal distance; Test type: Superiority or Other; p = 0.218, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 2: Comparison: Conventional Alar Base Cinch Suture; nasal height; Test type: Superiority or Other; p = 0.336, t-test, 2 sided; P- value < 0.05 was set as statistical significance
Statistical Analysis 3: Comparison: Conventional Alar Base Cinch Suture; Test type: Superiority or Other; p = 0.192, t-test, 2 sided; P- value < 0.05 was set as statistical significance
Statistical Analysis 4: Comparison: Conventional Alar Base Cinch Suture; nasal tip protrusion; Test type: Superiority or Other; p = 0.135, t-test, 2 sided; P value < 0.05 was set as statistical significance
Statistical Analysis 5: Comparison: Conventional Alar Base Cinch Suture; nasal width; Test type: Superiority or Other; p = 0.277, t-test, 2 sided; P value < 0.05 was set as statistical significance
Statistical Analysis 6: Comparison: Conventional Alar Base Cinch Suture; alar base width; Test type: Superiority or Other; p = 0.505, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 7: Comparison: Conventional Alar Base Cinch Suture; R nostril show vertical dimension; Test type: Superiority or Other; p = 0.299, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 8: Comparison: Conventional Alar Base Cinch Suture; L nostril show vertical dimension; Test type: Superiority or Other; p = 0.738, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 9: Comparison: Conventional Alar Base Cinch Suture; columellar length; Test type: Superiority or Other; p = 0.008, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 10: Comparison: Conventional Alar Base Cinch Suture; cutaneious height of upper lip; Test type: Superiority or Other; p = 0.116, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 11: Comparison: Conventional Alar Base Cinch Suture; overall upper lip height; Test type: Superiority or Other; p = 0.528, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 12: Comparison: Conventional Alar Base Cinch Suture; vermillion height of upper lip; Test type: Superiority or Other; p = 0.123, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 13: Comparison: Conventional Alar Base Cinch Suture; lower prolabial width; Test type: Superiority or Other; p = 0.250, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 14: Comparison: Conventional Alar Base Cinch Suture; upper lip protrusion; Test type: Superiority or Other; p = 0.706, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 15: Comparison: Modified Alar Cinch Suture; intercanthal distance; Test type: Superiority or Other; p = 0.804, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 16: Comparison: Modified Alar Cinch Suture; nasal height; Test type: Superiority or Other; p = 0.114, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 17: Comparison: Modified Alar Cinch Suture; Nasal length; Test type: Superiority or Other; p = 0.457, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 18: Comparison: Modified Alar Cinch Suture; Nasal tip protrusion; Test type: Superiority or Other; p = 0.565, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 19: Comparison: Modified Alar Cinch Suture; nasal width; Test type: Superiority or Other; p = 0.781, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 20: Comparison: Modified Alar Cinch Suture; alar base width; Test type: Superiority or Other; p = 0.164, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 21: Comparison: Modified Alar Cinch Suture; R nostril show vertical dimension; Test type: Superiority or Other; p = 0.554, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 22: Comparison: Modified Alar Cinch Suture; L nostril show vertical dimension; Test type: Superiority or Other; p = 0.508, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 23: Comparison: Modified Alar Cinch Suture; columellar length; Test type: Superiority or Other; p = 0.358, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 24: Comparison: Modified Alar Cinch Suture; cutaneous height of upper lip; Test type: Superiority or Other; p = 0.049, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 25: Comparison: Modified Alar Cinch Suture; overall upper lip height; Test type: Superiority or Other; p = 0.057, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 26: Comparison: Modified Alar Cinch Suture; vermillion height of upper lip; Test type: Superiority or Other; p = 0.062, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 27: Comparison: Modified Alar Cinch Suture; lower prolabial width; Test type: Superiority or Other; p = 0.029, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 28: Comparison: Modified Alar Cinch Suture; upper lip protrusion; Test type: Superiority or Other; p = 0.011, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 29: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; intercanthal distance; Test type: Superiority or Other; p = 0.211, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 30: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; nasal height; Test type: Superiority or Other; p = 0.102, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 31: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; nasal length; Test type: Superiority or Other; p = 0.136, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 32: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; nasal tip protrusion; Test type: Superiority or Other; p = 0.113, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 33: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; nasal width; Test type: Superiority or Other; p = 0.115, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 34: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; alar base width; Test type: Superiority or Other; p = 0.535, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 35: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; R nostril show vertical dimension; Test type: Superiority or Other; p = 0.850, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 36: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; L nostril show vertical dimension; Test type: Superiority or Other; p = 0.891, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 37: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; columellar length; Test type: Superiority or Other; p = 0.262, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 38: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; cutaneous height of upper lip; Test type: Superiority or Other; p = 0.344, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 39: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; overall upper lip height; Test type: Superiority or Other; p = 0.057, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 40: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; vermillion height of upper lip; Test type: Superiority or Other; p = 0.995, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 41: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; lower prolabial width; Test type: Superiority or Other; p = 0.440, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)
Statistical Analysis 42: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; upper lip protrusion; Test type: Superiority or Other; p = 0.078, t-test, 2 sided; P-value < 0.05 was set as statistical significance(*)

3. Secondary Outcome: 1 Nasolabial Angular Parameters
Description: 2D nasolabial angular parameter: Nasolabial angle (NLA) (The NLA was a two dimensional measurement and was measured at the midsagittal plane with Image J software®)
Time Frame: up to post-operation 6 months
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Modified Alar Cinch Suture | Conventional Alar Base Cinch Suture
Number analyzed (Participants) | 24 | 24
degree | 3.25 (7.25) | 2.92 (8.28)
Statistical Analysis 1: Comparison: Conventional Alar Base Cinch Suture; Test type: Superiority or Other; p = 0.104, t-test, 2 sided — intergroup difference of conventional group; P value < 0.05 was set as statistical significance
Statistical Analysis 2: Comparison: Modified Alar Cinch Suture; Test type: Superiority or Other; p = 0.043, t-test, 2 sided — Intergroup difference of modified group; P value <0.05 was set as statistical significance
Statistical Analysis 3: Comparison: Modified Alar Cinch Suture vs Conventional Alar Base Cinch Suture; Test type: Superiority or Other; p = 0.888, t-test, 2 sided; P value < 0.05 was set as statistical significance

ADVERSE EVENTS:
Time Frame: 6 months after surgery
Groups:
- Modified Alar Cinch Suture: modified extraoral alar cinch suture techniques suture from not only ANS and nasalis muscle, but also through the dermis layer of the alar base.
  modified extraoral alar base cinch technique: modified alar cinch suture technique performed after the maxillary Lefort I osteotomy.
- Conventional Alar Base Cinch Suture: conventional nasal cinch alar base technique: suture goes through bilateral alar base and anterior nasal spine(ANS) and nasalis muscle intra-orally
  conventional nasal alar cinch suture technique: conventional alar cinch suture technique performed after the maxillary Lefort I osteotomy.
Arm/Group | Modified Alar Cinch Suture | Conventional Alar Base Cinch Suture
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
no financial PI disclosure